CLINICAL TRIAL: NCT02016131
Title: Application of Color-coded Quantitative Digital Subtraction Angiography in Evaluation of Prognosis After Endovascular Repairment of Abdominal Aortic Aneurysm
Brief Title: CQDSA in Evaluation of Prognosis After EVAR
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Siemens Ltd., China, Shanghai, China. (Unknown)
Responsible Party: Principal Investigator, Zhenyu Shi, Associate Prof., Shanghai Zhongshan Hospital
Other Study IDs: CQDSA_EVAR
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2015-05

CONDITIONS: Endoleak; Aortic Aneurysm, Abdominal
Keywords: endoleak; EVAR; AAA; CQDSA
MeSH Terms: conditions — Endoleak; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- none endoleak events: Patients who have no further endoleaks related adverse events including aneurysm enlargement and rupture or persistent endoleaks.
- Endoleak events: Patients who undergo endoleaks related adverse events or persistent endoleaks during follow up.

SUMMARY:
Re-hospitalization or re-intervention is sometimes necessary to treat type I and type III endoleaks after EVAR for its persistent increasing of pressure in aneurysm lumen. Color-coded quantitative digital subtraction angiography (CQDSA) provides an easy and quick way to post-process the traditional digital subtraction angiography (DSA) which converts the peak time of the maximal contrast medium intensity into a single polychromatic image. With the help of CQDSA, a quantitative evaluation of the endoleak hemodynamics and a risk analysis of the type I or type III endoleak could be performed during the EVAR procedure. This approach may offer an objective assessment of the needs for immediate re-intervention, conservative therapy or treatment endpoint in the future.

DETAILED DESCRIPTION:
Intra-procedural DSA series are transferred to a research workstation to generate the color-coded images and make quantitative measurements. Region of interest (ROI) measurements are performed equivalently in the endoleak and the aorta after the image generation. There are three kinds of ROIs including a small circle area with the shortest time to peak, a circle area with peak contrast intensity and the whole endoleak area. The ROI and a reference at the same latitude within the aorta are selected to undergo measurement which reflected the endoleak hemodynamics of the endoleak to the utmost extent.

The following parameters will be acquired through the CQDSA for analysis.

1. Time-versus-ROI contrast intensity graph. The graph contains one endoleak ROI flow curve and one reference aortic flow curve (Ref). The x-axis shows time from 0 second to the maximum frame time of the image. The y-axis shows the sum of pixel intensities, namely total contrast, representing the contrast concentration within the ROI.
2. ROI Peak/Ref Peak. It is the ratio of intensity peak between the endoleak and the reference in the aorta.
3. ROI TTP (Time to peak). Peak time of ROI in the vicinity of endoleak entry.
4. ROI AUC/Ref AUC. Area under curve (AUC) is calculated through Time-versus-ROI contrast intensity graph. The parameter here is the ratio of ROI AUC in endoleak to the reference.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present type I or/and type III endoleak after EVAR for AAA and complete at least 3 months' follow up.

Exclusion Criteria:

* Patients who

  1. undergo surgeries which involve the segment covered by EVAR;
  2. present connective tissue disease, such as Marfan's Syndrome or vasculitis.
  3. present abdominal aortic dissection.
  4. present AAA rupture.
  5. die from non aneurysm-reltated reasons or are lost during follow up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present type I endoleak after EVAR for AAA.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time-versus-ROI contrast intensity graph. | 15 seconds
  The graph contains one endoleak ROI flow curve and one reference aortic flow curve (Ref). The x-axis shows time from 0 second to the maximum frame time of the image. The y-axis shows the sum of pixel intensities, namely total contrast, representing the contrast concentration within the ROI.
ROI Peak/Ref Peak | 15 seconds
  It is the ratio of intensity peak between the endoleak and the reference in the aorta.
ROI TTP (Time to peak) | 15 seconds
  Peak time of ROI in the vicinity of endoleak entry
ROI AUC/Ref AUC | 15 seconds
  Area under curve (AUC) is calculated through Time-versus-ROI contrast intensity graph. The parameter here is the ratio of ROI AUC in endoleak to the reference.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Fu, MD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China

REFERENCES:
- [Background] Lederle FA, Johnson GR, Wilson SE, Chute EP, Littooy FN, Bandyk D, Krupski WC, Barone GW, Acher CW, Ballard DJ. Prevalence and associations of abdominal aortic aneurysm detected through screening. Aneurysm Detection and Management (ADAM) Veterans Affairs Cooperative Study Group. Ann Intern Med. 1997 Mar 15;126(6):441-9. doi: 10.7326/0003-4819-126-6-199703150-00004. PMID 9072929
- [Background] Thompson AR, Cooper JA, Ashton HA, Hafez H. Growth rates of small abdominal aortic aneurysms correlate with clinical events. Br J Surg. 2010 Jan;97(1):37-44. doi: 10.1002/bjs.6779. PMID 20013940
- [Background] Brady AR, Thompson SG, Fowkes FG, Greenhalgh RM, Powell JT; UK Small Aneurysm Trial Participants. Abdominal aortic aneurysm expansion: risk factors and time intervals for surveillance. Circulation. 2004 Jul 6;110(1):16-21. doi: 10.1161/01.CIR.0000133279.07468.9F. Epub 2004 Jun 21. PMID 15210603
- [Background] Reed WW, Hallett JW Jr, Damiano MA, Ballard DJ. Learning from the last ultrasound. A population-based study of patients with abdominal aortic aneurysm. Arch Intern Med. 1997 Oct 13;157(18):2064-8. doi: 10.1001/archinte.157.18.2064. PMID 9382661
- [Background] Scott RA, Ashton HA, Lamparelli MJ, Harris GJ, Stevens JW. A 14-year experience with 6 cm as a criterion for surgical treatment of abdominal aortic aneurysm. Br J Surg. 1999 Oct;86(10):1317-21. doi: 10.1046/j.1365-2168.1999.01227.x. PMID 10540141
- [Background] Scott RA, Wilson NM, Ashton HA, Kay DN. Is surgery necessary for abdominal aortic aneurysm less than 6 cm in diameter? Lancet. 1993 Dec 4;342(8884):1395-6. doi: 10.1016/0140-6736(93)92756-j. PMID 7901685
- [Background] Mortality results for randomised controlled trial of early elective surgery or ultrasonographic surveillance for small abdominal aortic aneurysms. The UK Small Aneurysm Trial Participants. Lancet. 1998 Nov 21;352(9141):1649-55. PMID 9853436
- [Background] Lederle FA, Wilson SE, Johnson GR, Reinke DB, Littooy FN, Acher CW, Ballard DJ, Messina LM, Gordon IL, Chute EP, Krupski WC, Busuttil SJ, Barone GW, Sparks S, Graham LM, Rapp JH, Makaroun MS, Moneta GL, Cambria RA, Makhoul RG, Eton D, Ansel HJ, Freischlag JA, Bandyk D; Aneurysm Detection and Management Veterans Affairs Cooperative Study Group. Immediate repair compared with surveillance of small abdominal aortic aneurysms. N Engl J Med. 2002 May 9;346(19):1437-44. doi: 10.1056/NEJMoa012573. PMID 12000813
- [Background] Moll FL, Powell JT, Fraedrich G, Verzini F, Haulon S, Waltham M, van Herwaarden JA, Holt PJ, van Keulen JW, Rantner B, Schlosser FJ, Setacci F, Ricco JB; European Society for Vascular Surgery. Management of abdominal aortic aneurysms clinical practice guidelines of the European society for vascular surgery. Eur J Vasc Endovasc Surg. 2011 Jan;41 Suppl 1:S1-S58. doi: 10.1016/j.ejvs.2010.09.011. No abstract available. PMID 21215940
- [Background] Jens S, Marquering HA, Koelemay MJ, Reekers JA. Perfusion angiography of the foot in patients with critical limb ischemia: description of the technique. Cardiovasc Intervent Radiol. 2015 Feb;38(1):201-5. doi: 10.1007/s00270-014-1036-5. Epub 2014 Dec 13. PMID 25501266
- [Background] Benndorf G. Color-coded digital subtraction angiography: the end of a monochromatic era? AJNR Am J Neuroradiol. 2010 May;31(5):925-7. doi: 10.3174/ajnr.A2077. Epub 2010 Apr 15. No abstract available. PMID 20395396
- [Background] Mehndiratta A, Knopp MV, Zechmann CM, Owsijewitsch M, von Tengg-Kobligk H, Zamecnik P, Kauczor HU, Choyke PL, Giesel FL. Comparison of diagnostic quality and accuracy in color-coded versus gray-scale DCE-MR imaging display. Int J Comput Assist Radiol Surg. 2009 Sep;4(5):457-62. doi: 10.1007/s11548-009-0356-4. Epub 2009 Jun 4. PMID 20033528
- [Background] Tenjin H, Asakura F, Nakahara Y, Matsumoto K, Matsuo T, Urano F, Ueda S. Evaluation of intraaneurysmal blood velocity by time-density curve analysis and digital subtraction angiography. AJNR Am J Neuroradiol. 1998 Aug;19(7):1303-7. PMID 9726473
- [Background] Strother CM, Bender F, Deuerling-Zheng Y, Royalty K, Pulfer KA, Baumgart J, Zellerhoff M, Aagaard-Kienitz B, Niemann DB, Lindstrom ML. Parametric color coding of digital subtraction angiography. AJNR Am J Neuroradiol. 2010 May;31(5):919-24. doi: 10.3174/ajnr.A2020. Epub 2010 Feb 18. PMID 20167651
- [Background] Khanafer KM, Bull JL, Upchurch GR Jr, Berguer R. Turbulence significantly increases pressure and fluid shear stress in an aortic aneurysm model under resting and exercise flow conditions. Ann Vasc Surg. 2007 Jan;21(1):67-74. doi: 10.1016/j.avsg.2006.10.009. PMID 17349339
- [Background] Hunter GJ, Hunter JV, Brown NJ. Parametric imaging using digital subtraction angiography. Br J Radiol. 1986 Jan;59(697):7-11. doi: 10.1259/0007-1285-59-697-7. PMID 3512003
- [Background] Veith FJ, Baum RA, Ohki T, Amor M, Adiseshiah M, Blankensteijn JD, Buth J, Chuter TA, Fairman RM, Gilling-Smith G, Harris PL, Hodgson KJ, Hopkinson BR, Ivancev K, Katzen BT, Lawrence-Brown M, Meier GH, Malina M, Makaroun MS, Parodi JC, Richter GM, Rubin GD, Stelter WJ, White GH, White RA, Wisselink W, Zarins CK. Nature and significance of endoleaks and endotension: summary of opinions expressed at an international conference. J Vasc Surg. 2002 May;35(5):1029-35. doi: 10.1067/mva.2002.123095. PMID 12021724
- [Background] Hinnen JW, Koning OH, van Bockel JH, Hamming JF. Aneurysm sac pressure after EVAR: the role of endoleak. Eur J Vasc Endovasc Surg. 2007 Oct;34(4):432-41; discussion 442-3. doi: 10.1016/j.ejvs.2007.05.022. Epub 2007 Aug 1. PMID 17669670
- [Derived] Zhou M, Su Z, Shi Z, Fu W, Meng X, Wang Y, Guo B, Huang K. Application of color-coded quantitative digital subtraction angiography in predicting the outcomes of immediate type I and type III endoleaks. J Vasc Surg. 2017 Sep;66(3):760-767. doi: 10.1016/j.jvs.2016.11.048. Epub 2017 Feb 16. PMID 28216350